CLINICAL TRIAL: NCT01777438
Title: Evaluating Symptom Control in in Allergic Rhinitis at Three Years After Starting Immunotherapy
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: 102012
Record Dates: First submitted 2013-01-23; First posted 2013-01-28 (Estimated); Results first posted 2013-12-17 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-10

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- control group: a control group of AR patients who visited the ear nose and throat (ENT) department of the University Hospitals Leuven in the same time period
- patients having SCIT: patients who started immunotherapy at the Department of Allergology of the University Hospitals Leuven between November 2007 and February 2010.

SUMMARY:
Allergic rhinitis (AR) is defined as inflammation of the nasal mucosa after exposition to an allergen in sensitized patients. AR causes not only nasal symptoms such as sneezing, itchy nose, rhinorrhea and nasal obstruction, but also has a significant impact on quality of life. Symptom control and overall satisfaction in patients undergoing subcutaneous immunotherapy (SCIT) or sublingual immunotherapy (SLIT) on the long term has not yet been investigated so far.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with at least 2 AR symptoms and a positive skin prick test for the 20 most prevalent inhalant allergens (house dust mites, grass pollen, tree pollen, animal dander, Alternaria, Penicillium and Cladosporium) in Belgium.
2. Moderate/severe and/or persistent AR according to ARIA guidelines
3. Age > 18 and < 60 years.
4. Written informed consent
5. Dutch, French or English speaking patients

Exclusion Criteria:

Exclusion criteria

1. Age < 18 and > 60 years
2. Patients with mild AR
3. Patients not being able to give an informed consent
4. Patients being enrolled in other clinical trials
5. No knowledge of Dutch, French or English

Ages: 19 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients who started immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 434 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hellings, MD, Principal Investigator — UZ Leuven
Locations (2):
- Belgium (2):
  - ORL, Leuven, Vlaams-Brabant
  - UZ Leuven, Leuven, Vlaams-brabant

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: a control group of AR patients who visited the ENT department of the University Hospitals Leuven in the same time period
Period: Overall Study
Arm/Group | Control Group | Patients Having SCIT
Started | 352 | 82
Completed | 352 | 82
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Patients Having SCIT | Total
Number analyzed (Participants) | 352 | 82 | 434
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 352 | 82 | 434
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 201 | 48 | 249
  Male | 151 | 34 | 185
Region of Enrollment [Number; unit: participants]
  Belgium | 352 | 82 | 434

OUTCOME MEASURES:

1. Primary Outcome: Current Medication Use Three Years After Diagnosis of AR
Description: Percentage patients in both groups that still use medication for their allergic rhinitis symptoms, 3 years after starting their therapy (non IT-group vs IT-group)
Time Frame: 3 years after starting SCIT
Measure: Number; unit: percentage of participants
Arm/Group | Control Group | Patients Having SCIT
Number analyzed (Participants) | 352 | 82
percentage of participants | 61 | 29

2. Secondary Outcome: Percentage of Patients Having Controlled Allergic Rhinosinusitis (AR) Symptoms 3 Years After Starting Treatment
Description: Based on the proposed cut-off value of VAS < 5/10 for total nasal symptoms (TNS), rhinitis was considered as being controlled in 69 IT patients (84%) versus 223 (63%) non-IT patients
Time Frame: 3 years after starting SCIT
Measure: Number; unit: percentage of participants
Arm/Group | Control Group | Patients Having SCIT
Number analyzed (Participants) | 352 | 82
percentage of participants | 63 | 84

3. Primary Outcome: Degree of Symptom Control 3 Years After IT or 3 Years After Medical Treatment With VAS of Total Nasal Symptom < 5/10 Defined as a Controlled Situation.
Description: Visual analogue scale (VAS) scores for TNS experienced during the last 4 weeks. Visual analog scales (VAS) have been used to rate the presence of symptoms or impairment of the daily activities. Patients had to answer each question by indicating a position with a vertical line between two endpoints, 0 cm for not bothersome versus 10 cm for extremely bothersome. In this way each question is scored between 0 and 10 points.
Time Frame: 3 years after diagnosis
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control Group | Patients Having SCIT
Number analyzed (Participants) | 353 | 81
Score on a scale | 3.7 (2.8) | 2.5 (2.3)

4. Secondary Outcome: Percentage of Patients That Met ARIA Criteria for Mild AR Symtoms at a Mean Interval of 3 Years After Diagnosis
Description: ARIA classification of AR is made by duration and severity of AR symptoms. Here are calculated the number of patients having mild acute rhinitis.
  Clinical practice guidelines such as the Allergic Rhinitis and its Impact on Asthma (ARIA) document focus on the quality of life as a principal consideration in assessment and treatment of AR
Time Frame: 3 years after diagnosis
Measure: Number; unit: percentage of participants
Arm/Group | Control Group | Patients Having SCIT
Number analyzed (Participants) | 353 | 81
percentage of participants | 32 | 78

ADVERSE EVENTS:
Arm/Group | Control Group | Patients Having SCIT
Serious Adverse Events (participants affected / at risk) | 0/352 | 0/82
Other Adverse Events (participants affected / at risk) | 0/352 | 0/82

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes